CLINICAL TRIAL: NCT02965040
Title: A Phase 1 Study to Evaluate the Pharmacokinetics of Roxadustat in Subjects With Different Degrees of Renal Function
Brief Title: A Phase 1 Study of Roxadustat in Subjects With Different Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0543; 2015-002565-28 (EudraCT Number)
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Normal Renal Function; Impaired Renal Function
Keywords: ASP1517; Normal renal function; Dialysis; Roxadustat; Metabolites; Pharmacokinetics; Impaired renal function
MeSH Terms: conditions — Renal Insufficiency | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Roxadustat: subjects with normal renal function (Experimental): Normal renal function: eGFR is equal to or greater than 90 mL/min/1.73 m^2. Single dose of roxadustat
  Interventions: Drug: Roxadustat
- Roxadustat: subjects with severely impaired renal function (Experimental): Severely impaired renal function: eGFR is less than 30 mL/min/1.73 m^2. Single dose of roxadustat
  Interventions: Drug: Roxadustat
- Roxadustat: subjects with ESRD on CAPD or APD (Experimental): ESRD subjects on CAPD or APD need to be on the same mode of dialysis for at least 4 months. Single dose of roxadustat
  Interventions: Drug: Roxadustat
- Roxadustat: subjects with ESRD on HD or HDF (Experimental): ESRD subjects on HD or HDF need to be on the same mode of dialysis for at least 4 months and should have dialysis sessions three times weekly. Single dose of roxadustat, in both treatment periods
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Oral
  Other Names: FG-4592; ASP1517

SUMMARY:
For subjects with normal renal function or severely impaired renal function, this study will evaluate the pharmacokinetics of roxadustat and its main metabolites in plasma and urine.

For subjects with end stage renal disease (ESRD) on continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dialysis (APD), this study will evaluate the pharmacokinetics of roxadustat and its main metabolites in plasma, urine and dialysate.

For subjects with ESRD on hemodialysis (HD) or hemodiafiltration (HDF), this study will evaluate the pharmacokinetics of roxadustat and its main metabolites in plasma, urine and dialysate and also the effect of dialysis on the pharmacokinetics of roxadustat and its main metabolites.

DETAILED DESCRIPTION:
This is a phase 1, open-label study in two sites. There will be four different renal function groups.

For all subjects:

Subjects will be allocated to the normal and severely impaired renal function groups based on estimated glomerular filtration rate (eGFR), calculated with the abbreviated modification of diet in renal disease (MDRD) equation. The eGFR will be based on the serum creatinine concentration and is assessed at screening and at day -2. The eGFR obtained at screening will determine the allocation.

Subjects will be allocated to the ESRD groups based on their dialysis requirements.

Subjects with normal and severely impaired renal function, and subjects with ESRD on CAPD or APD:

Screening will take place from day -30 to day -3 and the subjects will be admitted to the clinical unit on day -2. The treatment period lasts 8 days, during which the subjects will receive a single oral dose of roxadustat in the morning of day 1 Subjects will complete the treatment period on day 6, provided that all required assessments have been performed and there are no medical reasons for a prolonged follow-up. The study will be completed with an end-of-study visit (ESV), which will take place between 5 and 9 days after the last treatment period-defined assessment (or after early withdrawal).

Subjects with ESRD on HD or HDF:

Screening will take place from day -30 to day -3 and subjects will complete 2 treatment periods of 8 days (period 1) and 7 days (period 2) in order to evaluate the pharmacokinetics of roxadustat with a single oral dose of roxadustat on day 1 of both periods after and before dialysis.

Subjects will complete the treatment period 1 on day 6 followed by a wash-out period which is minimally 1 week and maximally 3 weeks. Subjects will complete period 2 on day 6, provided that all required assessments have been performed and there are no medical reasons for a prolonged follow-up. The study will be completed with an end-of-study visit (ESV), which will take place between 5 and 9 days after the last treatment period-defined assessment (or after early withdrawal).

All subjects:

Safety assessments will be performed throughout the study. An optional biobanking sample may be taken for potential exploratory, retrospective, gene polymorphism analysis. Roxadustat plasma, urine, and dialysate samples will be stored for potential exploratory metabolic profiling or exploratory biomarker analysis after the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

* Subject has a body weight of 45 to 160 kg, inclusive.
* For subjects with ESRD on CAPD or APD body weight should be recorded as the measured body weight minus abdominal dialysis fluid based on the last filling. For subjects with ESRD on HD or HDF the post-dialysis body weight will be recorded.

Specific inclusion criteria for subjects with normal renal function:

* Subject is a healthy male or female subject aged 40 to 75 years, inclusive.
* Subject must have a pre-dose eGFR value based on the abbreviated MDRD method of greater than or equal to 90 mL/min/1.73 m^2.

Specific inclusion criteria for subjects with severely impaired renal function:

* Subject is a male or female subject aged 18 to 75 years, inclusive.
* Subject must have a pre-dose eGFR value based on the abbreviated MDRD method [screening] of <30 mL/min/1.73 m^2 and not be on dialysis.

Specific inclusion criteria for subjects with ESRD on CAPD or APD:

* Subject is a male or female subject aged 18 to 75 years, inclusive.
* Subject is on CAPD or APD treatment with the same mode of dialysis for at least 4 months prior to admission to the clinical unit.

Specific inclusion criteria for subjects with ESRD on HD or HDF:

* Subject is a male or female subject aged 18 to 75 years, inclusive.
* Subject is on HD or HDF treatment with the same mode of dialysis for at least 4 months prior to admission to the clinical unit and should have dialysis sessions three times weekly.

Specific inclusion criteria for subjects with impaired renal function including severly impaired renal function and ESRD:

* If a subject is being treated with short-acting ESAs, the subject agrees to discontinue treatment for at least 14 days prior to admission.

Exclusion Criteria:

Exclusion criteria for all subjects:

* Subject has a known or suspected hypersensitivity to Roxadustat or any components (e.g., lactose) of the formulations used.
* Subject has any clinically significant history of allergic conditions (including drug allergies or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG), and clinical study protocol-defined clinical laboratory tests at screening or day -2.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit.
* Subject has a history of drinking more than 21 units (male subjects) or more than 14 units (female subjects) of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit.
* Subject uses moderate or strong inducers of metabolism (e.g., barbiturates, rifampin) regularly in the 1 month prior to admission to the clinical unit.
* Subject must not consume grapefruit (or any grapefruit-containing products, including juice) or Seville oranges (or any Seville orange-containing products, including juice) within 7 days prior to admission to the clinical unit.
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), anti-hepatitis A virus (immunoglobulin M [IgM]), anti-hepatitis C virus, hepatitis B core antibody or anti-human immunodeficiency virus (HIV) type 1 or 2 [screening].
* Subject participated in any clinical study or has been treated with any investigational drugs within 28 days (or 5 half-lives whichever is longer), prior to screening.
* Subject has any condition which makes the subject unsuitable for clinical study participation.
* Subject is a vulnerable subject (e.g., subject kept in detention).

Specific exclusion criteria for subjects with normal renal function:

* Subjects aged greater than or equal to 40 and < 65:

  * Subject has a mean pulse < 45 or >90 bpm; mean systolic blood pressure <90 mmHg and >140 mmHg; mean diastolic blood pressure <50 mmHg and >90 mmHg at day -2. Vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically. If the mean pulse, systolic blood pressure or diastolic blood pressure exceeds the limits above, 1 additional triplicate can be taken [day -2].
* Subjects aged greater than or equal to 65 and less than or equal to 75:

  * Subject has a mean pulse <45 or >90 bpm; mean systolic blood pressure <90 mmHg and >160 mmHg; mean diastolic blood pressure <50 mmHg and >100 mmHg at day -2. Vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically. If the mean pulse, systolic blood pressure or diastolic blood pressure exceeds the limits above, 1 additional triplicate can be taken [day -2].
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, psychiatric, dermatologic, renal and/or other major disease or malignancy.
* Subjects aged greater than or equal to 40 and <65:

  * Subject has a mean corrected QT interval using Fridericia's formula (QTcF) >430 ms (for males) and >450 ms (for females) at day 2. If the mean QTcF exceeds the limits above, 1 additional triplicate Electrocardiogram (ECG) can be taken (day -2).
* Subjects aged greater than or equal to 65 and less than or equal to 75:

  * Subject has a mean QTcF >450 ms (for males) and >470 ms (for females) at day 2. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken (day -2).
* Subject has any of the liver chemistry tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT] and total bilirubin [TBL]) above 1.5 times the upper limit of normal (ULN) at day -2. In such a case, the assessment may be repeated once [day -2].
* Subject uses any prescribed or non-prescribed drugs (including vitamins, calcium, magnesium and iron supplements, natural- and herbal- remedies, e.g., St. John's Wort) within 2 weeks (or 5 half-lives, whichever is longer) prior to admission to the clinical unit, except for occasional use of paracetamol (up to 2 g per day) and oral contraceptives or hormone replacement therapy.

Specific exclusion criteria for subjects with impaired renal function (including severely impaired renal function and ESRD):

* Subject has a mean pulse <45 or >90 bpm; mean systolic blood pressure <90 mmHg and >160 mmHg; mean diastolic blood pressure <50 mmHg and >100 mmHg at day -2. Vital signs measurements, taken in triplicate after the subject has been resting in supine position for 5 minutes; pulse will be measured automatically. If the mean pulse, systolic blood pressure or diastolic blood pressure exceeds the limits above, 1 additional triplicate can be taken [day -2].
* Subject has a history of any clinically significant illness (other than renal disease and conditions related to the renal disease, such as stable diabetes and stable hypertension), medical condition, or laboratory abnormality within 3 months prior to screening that would preclude participation in the clinical study.
* Subject has used immunosuppressant drugs or drugs used to treat malignancies (including corticosteroids at doses >10 mg prednisolone per day or equivalent) within 3 months prior to admission to the clinical unit.
* Subject is anticipated to undergo surgery that is expected to lead to significant blood loss during the clinical study period or anticipated coronary revascularization.
* Subject has an anticipated use of the following prohibited medication during the treatment and/or follow-up of the study:

  * Oral multivalent cation-containing drugs and mineral supplements (e.g., iron, calcium, magnesium, aluminium), anion-exchange resins (e.g., colestyramine), sucralfate or magnesium- or aluminium-containing antacids, phosphate binders, and iron-chelating agents are not allowed from 24 hours before until 48 hours after dosing.
  * Short-acting intravenous (IV) or subcutaneous (SC) Erythropoiesis stimulating agents (ESA) are not allowed within 2 weeks prior to admission to the clinical unit until the ESV.
  * Dapsone in any dose amount or anticipated chronic use of paracetamol >2 g/day or nonsteroidal anti-inflammatory drugs (NSAIDs), except for low dose aspirin/acetylsalicylic acid, is not allowed from admission to the clinical unit until the ESV.
* Subject has not been on a stable dose of concomitant medication to treat concurrent chronic conditions for at least 2 weeks (or 5 half-lives of the drug, whichever is longer) prior to admission to the clinical unit (minor dose changes are allowed in agreement with Sponsor). Doses of statins should not exceed the capped maximum daily doses at admission to the clinical unit. Rosuvastatin use is not allowed.
* Subject who requires, or is likely to require, any new concomitant medication from the time of screening until the ESV.
* Subject has used any non-essential prescribed and non-prescribed drugs (including vitamins, natural- and herbal-remedies (e.g., St. John's Wort) within 2 weeks (or 5 half-lives, whichever is longer) prior to admission to the clinical unit.
* Subject has a mean QTcF >450 ms (for males) and >470 ms (for females) at day 2. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken (day -2).
* Subject who has renal disease secondary to malignancy.
* Subject who has a fluctuating or rapidly deteriorating renal function within 4 weeks prior to admission to the clinical unit, as indicated by strongly varying or worsening of clinical and/or laboratory signs of renal impairment within the screening period.
* Subject with serum uric acid >2 x the ULN. In such a case the assessment may be repeated once [day -2].
* Subject with any of the liver chemistry tests (AST, ALT and TBL) out of range as indicated below. In such a case the assessment may be repeated once [day -2].

  * ALT or AST >3 x ULN
  * TBL >1.5 x ULN
* Subject has had any prior organ transplant (that has not been explanted) or subject is scheduled for organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Roxadustat in plasma: Cmax | Up to day 6
  Cmax: Maximum concentration
Pharmacokinetics of Roxadustat in plasma: Cmax,u | Up to day 6
  Cmax,u: Maximum concentration of unbound compound
Pharmacokinetics of Roxadustat in plasma: AUCinf | Up to day 6
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
Pharmacokinetics of Roxadustat in plasma: AUCinf,u | Up to day 6
  AUCinf,u: Area under the concentration-time curve from the time of dosing extrapolated to time infinity for unbound concentration
Pharmacokinetics of Roxadustat in plasma: AUClast | Up to day 6
  AUClast: Area under the concentration-time curve from the time of dosing to the last measurable concentration (Clast)
Pharmacokinetics of Roxadustat in plasma: AUClast,u | Up to day 6
  AUClast,u: Area under the concentration-time curve from the time of dosing to the last measurable concentration (Clast) for unbound concentration
Pharmacokinetics of Roxadustat in plasma: CL/F | Up to day 6
  CL/F: Apparent total systemic clearance after single or multiple extravascular dosing
Pharmacokinetics of Roxadustat in plasma: CLu/F | Up to day 6
  CLu/F: Apparent total systemic clearance of unbound compound after extravascular dosing
Pharmacokinetics of Roxadustat in plasma: fu | Up to day 6
  fu: Fraction of parent or metabolite available systemically unbound (= free fraction)
Pharmacokinetics of Roxadustat in plasma: tmax | Up to day 6
  tmax: Time of the maximum concentration
Pharmacokinetics of Roxadustat in plasma t1/2 | Up to day 6
  t1/2: Terminal elimination half-life
Pharmacokinetics of Roxadustat in plasma: Vz/F | Up to day 6
  Vz/F: Apparent volume of distribution during the terminal elimination phase after single extravascular dosing
Pharmacokinetics of Roxadustat in plasma: Vz,u/F | Up to day 6
  Vz,u/F: Apparent volume of distribution during the terminal elimination phase of unbound compound after extravascular dosing
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: Cmax | Up to day 6
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: AUCinf | Up to day 6
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: AUClast | Up to day 6
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: tlag | Up to day 6
  tlag: Time prior to the time corresponding to the first measurable (non-zero) concentration
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: tmax | Up to day 6
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: t1/2 | Up to day 6
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: MPR | Up to day 6
  MPR: Metabolite to parent ratio of AUC using AUC (corrected) for the metabolite (corrected by molecular weight ratio of parent to metabolite)
Pharmacokinetics of O-glucoside -Roxadustat in plasma: Cmax | Up to day 6
Pharmacokinetics of O-glucoside-Roxadustat in plasma: AUCinf | Up to day 6
Pharmacokinetics of O-glucoside-Roxadustat in plasma: AUClast | Up to day 6
Pharmacokinetics of O-glucoside-Roxadustat in plasma: tlag | Up to day 6
  tlag: Time prior to the time corresponding to the first measurable (non-zero) concentration
Pharmacokinetics of O-glucoside-Roxadustat in plasma: tmax | Up to day 6
Pharmacokinetics of O-glucoside-Roxadustat in plasma: t1/2 | Up to day 6
Pharmacokinetics of O-glucoside-Roxadustat in plasma: MPR | Up to day 6
  MPR: Metabolite to parent ratio of AUC using AUC(corrected) for the metabolite (corrected by molecular weight ratio of parent to metabolite)
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: Cmax | Up to day 6
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: AUCinf | Up to day 6
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: AUClast | Up to day 6
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: tlag | Up to day 6
  tlag: Time prior to the time corresponding to the first measurable (non-zero) concentration
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: tmax | Up to day 6
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: t1/2 | Up to day 6
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: MPR | Up to day 6
Pharmacokinetics of Roxadustat in urine: CLR | Up to day 4
  CLR: Renal clearance
Pharmacokinetics of Roxadustat in urine: CLR,u | Up to day 4
  CLR,u: Renal clearance of unbound drug
Pharmacokinetics of Roxadustat in urine: Aeinf | Up to day 4
  Aeinf: Cumulative amount of compound excreted into urine from time of dosing extrapolated to time infinity
Pharmacokinetics of Roxadustat in urine: Aeinf% | Up to day 4
  Aeinf%: Percent of drug dose excreted into urine (Aeinf) from time of dosing extrapolated to time infinity
Pharmacokinetics of Roxadustat in urine: Aelast | Up to day 4
  Aelast: Cumulative amount of drug excreted into urine from time of dosing up to the collection time of the last measurable concentration
Pharmacokinetics of Roxadustat in urine: Aelast% | Up to day 4
  Aelast%: Percent of drug dose excreted into urine (Aelast) from time of dosing up to the collection time of the last measurable concentration
Pharmacokinetics of O-glucuronide-Roxadustat in urine: CLR | Up to day 4
Pharmacokinetics of O-glucuronide-Roxadustat in urine: Aeinf | Up to day 4
Pharmacokinetics of O-glucuronide-Roxadustat in urine: Aelast | Up to day 4
Pharmacokinetics of O-glucuronide-Roxadustat in urine: MPR based on Aeinf | Up to day 4
Pharmacokinetics of O-glucoside-Roxadustat in urine: CLR | Up to day 4
Pharmacokinetics of O-glucoside-Roxadustat in urine: Aeinf | Up to day 4
Pharmacokinetics of O-glucoside-Roxadustat in urine: Aelast | Up to day 4
Pharmacokinetics of O-glucoside-Roxadustat in urine: MPR based on Aeinf | Up to day 4
Pharmacokinetics of sulfate of hydroxy-Roxadustat in urine: CLR | Up to day 4
Pharmacokinetics of sulfate of hydroxy-Roxadustat in urine: Aeinf | Up to day 4
Pharmacokinetics of sulfate of hydroxy-Roxadustat in urine: Aelast | Up to day 4
Pharmacokinetics of sulfate of hydroxy-Roxadustat in urine: MPR based on Aeinf | Up to day 4
Pharmacokinetics of Roxadustat and its main metabolites in dialysate fluid: CLD | Up to day 2
  CLD: dialysis clearance. For ESRD subjects on CAPD or APD and for ESRD subjects on HD or HDF (treatment period 2 only)
Pharmacokinetics of Roxadustat in dialysate fluid: fD | Up to day 2
  fD: fraction of dose cleared by dialysis. For ESRD subjects on CAPD or APD and for ESRD subjects on HD or HDF (treatment period 2 only)
Pharmacokinetics of O-glucuronide-Roxadustat in urine: Aeinf% | Up to day 4
Pharmacokinetics of O-glucoside-Roxadustat in urine: Aeinf% | Up to day 4
Pharmacokinetics of sulfate of hydroxy-Roxadustat in urine: Aeinf% | Up to day 4
Pharmacokinetics of Roxadustat in plasma: Effective t½ 48 hours | Up to day 6
  Effective t½ 48 hours: Effective half-life based on a dosing interval of 48 hours
Pharmacokinetics of Roxadustat in plasma: Effective t½ 56 hours | Up to day 6
  Effective t½ 56 hours: Effective half-life based on a dosing interval of 56 hours
Pharmacokinetics of O-glucuronide-Roxadustat in plasma: TER | Up to day 6
  TER: Total exposure ratio
Pharmacokinetics of O-glucoside-Roxadustat in plasma: TER | Up to day 6
Pharmacokinetics of sulfate of hydroxy-Roxadustat in plasma: TER | Up to day 6

SECONDARY OUTCOMES:
Pharmacodynamics of Roxadustat assessed by measuring erythropoietin (EPO): Emax | Up to day 6
  Emax: Maximum effect
Pharmacodynamics of Roxadustat assessed by measuring erythropoietin (EPO): Emax-baseline | U to day 6
  Emax-baseline: Maximum effect from baseline
Pharmacodynamics of Roxadustat assessed by measuring erythropoietin (EPO): AUCE,last | Up to day 6
  AUCE,last: Area under the effect-time curve from the time of dosing to the last measurable effect
Pharmacodynamics of Roxadustat assessed by measuring erythropoietin (EPO): AUCE,last (baseline-corrected) | Up to day 6
  AUCE,last (baseline-corrected): Area under the effect-time curve from the time of dosing to the last measurable effect baseline corrected
Pharmacodynamics of Roxadustat assessed by measuring erythropoietin (EPO): tmax, EPO | Up to day 6
  tmax, EPO: Time to maximum EPO concentration
Safety assessed by nature, frequency, and severity of Adverse Events (AEs) | Up to End of Study (EOS) (Up to day 15, period 2)
Number of participants with vital signs abnormalities and/or adverse events related to treatment | Up to EOS (Up to day 15, period 2)
  Vital signs include: blood pressure (systolic and diastolic) and pulse
Safety assessed by routine 12- lead electrocardiogram (ECG) | Up to EOS (Up to day 15, period 2)
  Routine 12-lead ECG measurements will be performed for the different renal function groups, as applicable, after the subject has been in a supine position for at least 5 minutes. All routine 12-lead ECG data will be listed by subject
Safety assessed by continuous heart rate (HR) measurement | Up to day 2 (period 1)
  Holter
Number of participants with laboratory value abnormalities and/or adverse events related to treatment | Up to EOS (Up to day 15, period 2)
  Safety laboratory tests include: hematology, biochemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Chair — Astellas Pharma Europe B.V.
Locations (2):
- Site DE49001, München, Germany
- Site GB44001, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Studies conducted with product indications or formulations that remain in development are assessed after study completion to determine if Individual Participant Data can be shared. The plan to share Individual Participant Data is based on the status of product approval or termination of the compound, in addition to other study-specific criteria described on www.clinicalstudydatarequest.com under "Sponsor Specific Details for Astellas."

REFERENCES:
- [Derived] Groenendaal-van de Meent D, Kerbusch V, Kaspera R, Barroso-Fernandez B, Galletti P, Klein GK, den Adel M. Effect of Kidney Function and Dialysis on the Pharmacokinetics and Pharmacodynamics of Roxadustat, an Oral Hypoxia-Inducible Factor Prolyl Hydroxylase Inhibitor. Eur J Drug Metab Pharmacokinet. 2021 Jan;46(1):141-153. doi: 10.1007/s13318-020-00658-w. PMID 33165773
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=346